CLINICAL TRIAL: NCT03713593
Title: A Phase 3 Multicenter, Randomized, Double-blinded, Active-controlled, Clinical Study to Evaluate the Safety and Efficacy of Lenvatinib (E7080/MK-7902) in Combination With Pembrolizumab (MK-3475) Versus Lenvatinib in First-line Therapy of Participants With Advanced Hepatocellular Carcinoma (LEAP-002)
Brief Title: Safety and Efficacy of Lenvatinib (E7080/MK-7902) in Combination With Pembrolizumab (MK-3475) Versus Lenvatinib as First-line Therapy in Participants With Advanced Hepatocellular Carcinoma (MK-7902-002/E7080-G000-311/LEAP-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7902-002; MK-7902-002 (Other: MSD Protocol Number); E7080-G000-311 (Other: Eisai Protocol Number); LEAP-002 (Other: MSD); 194590 (Registry Identifier: JAPIC-CTI); 2018-002983-26 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: receptor tyrosine kinase inhibitor; programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lenvatinib plus pembrolizumab (Experimental): Participants receive lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Lenvatinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: lenvatinib; Biological: pembrolizumab
- lenvatinib plus placebo (Active Comparator): Participants receive lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally QD plus saline placebo by IV infusion on Day 1 Q3W. Saline placebo will be administered for up to 35 cycles (approximately 24 months). Lenvatinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: lenvatinib; Drug: saline placebo

INTERVENTIONS:
Drug: lenvatinib — Administered orally once a day
  Other Names: MK-7902; E7080; LENVIMA®
Biological: pembrolizumab — Administered as an IV infusion on Day 1 Q3W
  Other Names: MK-3475; KEYTRUDA®
  Arms: lenvatinib plus pembrolizumab
Drug: saline placebo — Administered as an IV infusion on Day 1 Q3W
  Arms: lenvatinib plus placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of lenvatinib (E7080/MK-7902) in combination with pembrolizumab (MK-3745) versus lenvatinib in combination with placebo as first-line therapy for the treatment of advanced hepatocellular carcinoma in adult participants.

The primary hypotheses of this study are that lenvatinib plus pembrolizumab is superior to lenvatinib plus placebo with respect to progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and ≥18 years of age at the time of signing the informed consent
* Has a diagnosis of hepatocellular carcinoma confirmed by radiology, histology, or cytology
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Has a Child-Pugh class A liver score
* Has a predicted life expectancy of >3 months
* Has at least one measurable hepatocellular carcinoma (HCC) lesion based on RECIST 1.1 as confirmed by BICR
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1
* Participants with hepatitis B will be eligible as long as their virus is well controlled

Exclusion Criteria:

* Has had esophageal or gastric variceal bleeding within the last 6 months
* Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* Has a preexisting Grade ≥3 gastrointestinal or non-gastrointestinal fistula
* Has clinically significant hemoptysis from any source or tumor bleeding within 2 weeks prior to the first dose of study intervention
* Has significant cardiovascular impairment within 12 months of the first dose of study intervention such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident stroke, or cardiac arrhythmia associated with hemodynamic instability
* Has had major surgery to the liver within 4 weeks prior to the first dose of study intervention
* Has had a minor surgery (ie, simple excision) within 7 days prior to the first dose of study intervention
* Has serious non-healing wound, ulcer, or bone fracture
* Has received any systemic chemotherapy for HCC or chemotherapy for any malignancy in the past 3 years
* Has received prior therapy with an anti-programmed cell death 1 (ant-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti- programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, or CD137)
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exceptions of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that has undergone potentially curative therapy
* Has a known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis as assessed by local site investigator
* Has severe hypersensitivity (≥Grade 3) to study intervention and/or any of their excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has urine protein ≥1 grams/24 hours
* Prolongation of corrected QT (QTc) interval to >480 milliseconds (corrected by Fridericia Formula)
* Has left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
* Has an active infection requiring systemic therapy with the exceptions of hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Has a known history of human immunodeficiency virus (HIV) infection
* Has known active tuberculosis (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (172):
- United States (21):
  - The University of Arizona Cancer Center - North Campus ( Site 0621), Tucson, Arizona
  - City of Hope Comprehensive Cancer Center ( Site 0587), Duarte, California
  - Scripps Health ( Site 0644), La Jolla, California
  - Pacific Hematology Oncology Associates ( Site 0588), San Francisco, California
  - UCLA ( Site 0589), Santa Monica, California
  - Georgetown University ( Site 0594), Washington D.C., District of Columbia
  - University of Miami, Sylvester Comprehensive Cancer Center ( Site 0596), Miami, Florida
  - Advent Health ( Site 0595), Orlando, Florida
  - Tampa General Medical Group ( Site 0629), Tampa, Florida
  - Emory University Winship Cancer Institute ( Site 0639), Atlanta, Georgia
  - University of Kansas Cancer Center ( Site 0600), Westwood, Kansas
  - Massachusetts General Hospital ( Site 0603), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 0716), Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai ( Site 0611), New York, New York
  - University of Rochester ( Site 0613), Rochester, New York
  - Stony Brook University Medical Center - Cancer Center ( Site 0612), Stony Brook, New York
  - University of Oklahoma Health Science Center ( Site 0625), Oklahoma City, Oklahoma
  - Oregon Health & Science University ( Site 0645), Portland, Oregon
  - Eastern Regional Medical Center, Inc. ( Site 0626), Philadelphia, Pennsylvania
  - Central Texas Veterans Healthcare System ( Site 0617), Temple, Texas
  - Cancer Care Northwest ( Site 0636), Spokane, Washington
- Australia (5):
  - Royal Prince Alfred Hospital ( Site 0001), Camperdown, New South Wales
  - Princess Alexandra Hospital ( Site 0007), Wooloongabba, Queensland
  - Monash Health-Monash Medical Centre ( Site 0004), Clayton, Victoria
  - St Vincents Hospital Melbourne ( Site 0003), Fitzroy, Victoria
  - Liverpool Hospital. ( Site 0002), Liverpool
- Canada (5):
  - BC Cancer-Vancouver Center ( Site 0056), Vancouver, British Columbia
  - London Health Sciences Centre ( Site 0053), London, Ontario
  - Sunnybrook Research Institute ( Site 0055), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0050), Toronto, Ontario
  - McGill University Health Centre ( Site 0052), Montreal, Quebec
- Chile (4):
  - Clinica Universidad Catolica del Maule ( Site 0065), Talca, Maule Region
  - Fundacion Arturo Lopez Perez ( Site 0064), Santiago, Santiago Metropolitan
  - Pontificia Universidad Catolica de Chile ( Site 0070), Santiago, Santiago Metropolitan
  - Instituto Clinico Oncologico del Sur ( Site 0067), Temuco
- China (19):
  - First Affiliated Hospital of Anhui Medical University ( Site 0095), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 0100), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0088), Beijing, Beijing Municipality
  - 900 Hospital of the Joint ( Site 0091), Fuzhou, Fujian
  - Guangdong General Hospital ( Site 0092), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0102), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0089), Harbin, Heilongjiang
  - Wuhan Union hospital Cancer Center ( Site 0105), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0094), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 0093), Changsha, Hunan
  - The 81st Hospital of PLA ( Site 0085), Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center ( Site 0086), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0090), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0087), Chengdu, Sichuan
  - Affiliated Tumor Hospital of Xinjiang Medical University ( Site 0109), Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University ( Site 0097), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 0110), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0101), Hangzhou, Zhejiang
  - Zhongshan Hospital Fudan University ( Site 0096), Shanghai
- Colombia (8):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0141), Medellín, Antioquia
  - Hospital Pablo Tobon Uribe ( Site 0144), Medellín, Antioquia
  - Hospital General de Medellin Luz Castro de Gutierrez ( Site 0137), Medellín, Antioquia
  - Biomelab S A S ( Site 0145), Barranquilla, Atlántico
  - Administradora Country SA - Clinica del Country ( Site 0146), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia E.S.E ( Site 0142), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 0140), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0139), Cali, Valle del Cauca Department
- France (9):
  - Institut Sainte Catherine ( Site 0167), Avignon
  - Hopital Beaujon ( Site 0160), Clichy
  - CHU Henri Mondor ( Site 0162), Créteil
  - CHRU de Lille - Hopital Claude Huriez ( Site 0159), Lille
  - Hopital de la Croix Rousse ( Site 0157), Lyon
  - Hopital Saint Joseph ( Site 0166), Marseille
  - Centre Hospitalier Regional du Orleans ( Site 0169), Orléans
  - Centre Eugene Marquis ( Site 0158), Rennes
  - CHU de Nancy Hopital Brabois Adultes ( Site 0164), Vandœuvre-lès-Nancy
- Germany (10):
  - Klinikum der Universitaet Aachen - RWTH ( Site 0185), Aachen
  - Universitaetsklinik Koeln ( Site 0189), Cologne
  - Universitaetsklinikum Carl Gustav Carus der TU Dresden ( Site 0178), Dresden
  - Universitaetsklinikum Essen ( Site 0188), Essen
  - Universitaetsklinikum Frankfurt ( Site 0180), Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0184), Hamburg
  - Universitaetsklinikum Leipzig ( Site 0187), Leipzig
  - Otto-Von-Guericke-Universitaet Magdeburg ( Site 0182), Magdeburg
  - Universitaetsklinikum Tuebingen ( Site 0179), Tübingen
  - Universitaetsklinikum Wuerzburg ( Site 0186), Würzburg
- Ireland (2):
  - St Vincents University Hospital ( Site 0242), Dublin
  - Mater Misericordiae University Hospital ( Site 0241), Dublin
- Italy (8):
  - Ospedale Sacro Cuore - Don Calabria ( Site 0289), Negrar, VR
  - Centro di Riferimento Oncologico de Aviano Istituto Nazionale Tumori ( Site 0292), Aviano
  - Policlinico S. Orsola-Malpighi ( Site 0286), Bologna
  - Istituto Oncologico Veneto ( Site 0287), Padua
  - Az Osp Univ Policlin Paolo Giaccone ( Site 0284), Palermo
  - Fondazione Salvatore Maugeri IRCCS. ( Site 0290), Pavia
  - Azienda Ospedaliero-Univers. Pisana Ospedale S. Chiara ( Site 0291), Pisa
  - Policlinico Universitario Campus Biomedico ( Site 0288), Roma
- Japan (22):
  - Aichi Cancer Center Hospital ( Site 0316), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0306), Kashiwa, Chiba
  - Kurume University Hospital ( Site 0322), Kurume, Fukuoka
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital ( Site 0304), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 0315), Kanazawa, Ishikawa-ken
  - Kagawa University Hospital ( Site 0324), Kita-gun, Kagawa-ken
  - Kagawa Prefectural Central Hospital ( Site 0325), Takamatsu, Kagawa-ken
  - Toranomon Hospital Kajigaya ( Site 0312), Kawasaki, Kanagawa
  - Yokohama City University Medical Center ( Site 0313), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 0314), Yokohama, Kanagawa
  - Kindai University Hospital ( Site 0319), Sayama, Osaka
  - Kyorin University Hospital ( Site 0309), Mitaka, Tokyo
  - Musashino Red Cross Hospital ( Site 0310), Musashino, Tokyo
  - Chiba University Hospital ( Site 0305), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 0321), Fukuoka
  - Hiroshima University Hospital ( Site 0320), Hiroshima
  - Osaka Red Cross Hospital ( Site 0317), Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 0323), Saga
  - National Cancer Center Hospital ( Site 0307), Tokyo
  - Toranomon Hospital ( Site 0311), Tokyo
  - The University of Tokyo Hospital ( Site 0308), Tokyo
  - Wakayama Medical University Hospital ( Site 0318), Wakayama
- Mexico (7):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0365), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0363), Mexico City, Mexico City
  - Centro de Investigacion Medica Aguascalientes ( Site 0355), Aguascalientes
  - CRYPTEX Investigacion Clinica S.A. de C.V. ( Site 0362), Mexico City
  - Medical Care and Research S.A. de C.V. ( Site 0359), Mérida
  - Oaxaca Site Management Organization S.C. ( Site 0366), Oaxaca City
  - Unidad Medica Oncologica ( Site 0369), Puebla City
- New Zealand (2):
  - Auckland City Hospital ( Site 0376), Auckland
  - Christchurch Hospital ( Site 0377), Christchurch
- Poland (6):
  - Wojewodzki Szpital Specjalistyczny nr 4 w Bytomiu ( Site 0419), Bytom, Silesian Voivodeship
  - Szpital Wojewodzki w Koszalinie im. Mikolaja Kopernika ( Site 0421), Koszalin, West Pomeranian Voivodeship
  - ID Clinic ( Site 0431), Mysłowice
  - Ars Medical Sp. z o.o. ( Site 0433), Piła
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0418), Warsaw
  - MTZ Clinical Research Sp. z o. o. ( Site 0427), Warsaw
- Russia (6):
  - N.N. Blokhin NMRCO ( Site 0439), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 0453), Moscow, Moscow
  - Railway Hospital of OJSC ( Site 0447), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 0446), Saint Petersburg, Sankt-Peterburg
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0450), Krasnoyarsk
  - Pyatigorsk Oncology Dispensary ( Site 0441), Pyatigorsk
- South Korea (5):
  - Seoul National University Bundang Hospital ( Site 0464), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 0462), Seoul, Seoul-teukbyeolsi [Seoul]
  - Yonsei University Severance Hospital ( Site 0463), Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center ( Site 0460), Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center ( Site 0461), Seoul
- Spain (8):
  - Hospital Universitari Vall d Hebron ( Site 0508), Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Puerta de Hierro ( Site 0513), Majadahonda, Madrid
  - Hospital General Universitario Gregorio Maranon ( Site 0504), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 0514), Madrid
  - Hospital Universitario La Paz ( Site 0510), Madrid
  - Complejo Hospitalario Universitario de Santiago ( Site 0506), Santiago de Compostela
  - Hospital Universitario Virgen del Rocio ( Site 0509), Seville
  - Hospital Universitario y Politecnico La Fe de Valencia ( Site 0505), Valencia
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 0529), Kaoshiung
  - China Medical University Hospital ( Site 0527), Taichung
  - Taichung Veterans General Hospital ( Site 0526), Taichung
  - National Cheng Kung University Hospital ( Site 0528), Tainan
  - National Taiwan University Hospital ( Site 0523), Taipei
  - Taipei Veterans General Hospital ( Site 0524), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0525), Taoyuan District
- Thailand (3):
  - Siriraj Hospital. Mahidol Univerisity ( Site 0213), Bangkok Noi, Bangkok
  - Songklanagarind Hospital ( Site 0214), Hat Yai, Changwat Songkhla
  - Chiang Mai University Maharaj Nakorn Chiang Mai Hospital ( Site 0211), Chiang Mai
- Turkey (Türkiye) (9):
  - Adana Sehir Hastanesi ( Site 0549), Adana
  - Hacettepe Uni. Tip Fakultesi ( Site 0553), Ankara
  - Abdurrahman Yurtaslan Onkoloji Hastanesi ( Site 0551), Ankara
  - Akdeniz Universitesi Tip Fakultesi ( Site 0548), Antalya
  - Trakya Universitesi Tip Fakultesi ( Site 0544), Edirne
  - Erzurum Ataturk University Faculty of Medicine ( Site 0546), Erzurum
  - Bezmi Alem Universitesi Tıp Fakultesi ( Site 0547), Istanbul
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi ( Site 0550), Konya
  - Inonu Universitesi Medical Fakultesi ( Site 0545), Malatya
- United Kingdom (6):
  - Royal Free London NHS Foundation Trust ( Site 0567), London, London, City of
  - Kings College Hospital NHS Foundation Trust ( Site 0565), London, London, City of
  - The Clatterbridge Cancer Centre NHS Foundation Trust ( Site 0573), Birkenhead
  - The Beatson West of Scotland Cancer Centre ( Site 0566), Glasgow
  - The Christie NHS Foundation Trust ( Site 0575), Manchester
  - Nottingham University Hospitals NHS Trust ( Site 0569), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Llovet JM, Kudo M, Merle P, Meyer T, Qin S, Ikeda M, Xu R, Edeline J, Ryoo BY, Ren Z, Masi G, Kwiatkowski M, Lim HY, Kim JH, Breder V, Kumada H, Cheng AL, Galle PR, Kaneko S, Wang A, Mody K, Dutcus C, Dubrovsky L, Siegel AB, Finn RS; LEAP-002 Investigators. Lenvatinib plus pembrolizumab versus lenvatinib plus placebo for advanced hepatocellular carcinoma (LEAP-002): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Dec;24(12):1399-1410. doi: 10.1016/S1470-2045(23)00469-2. PMID 38039993
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26856&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a radiologically, histologically- or cytologically-confirmed diagnosis of hepatocellular carcinoma (HCC) were recruited into this study.
Groups:
- Lenvatinib + Pembrolizumab: Participants received lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab was administered for up to 35 cycles (approximately 24 months). Lenvatinib was administered until progressive disease or unacceptable toxicity.
- Lenvatinib + Placebo: Participants received lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally QD plus saline placebo by IV infusion on Day 1 Q3W. Saline placebo was administered for up to 35 cycles (approximately 24 months). Lenvatinib was administered until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Started | 395 | 399
Completed | 0 | 0
Not Completed | 395 | 399
Not completed — Sponsor Decision | 73 | 41
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 314 | 349
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo | Total
Number analyzed (Participants) | 395 | 399 | 794
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (10.9) | 64.1 (12.1) | 64.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 72 | 150
  Male | 317 | 327 | 644
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 41 | 89
  Not Hispanic or Latino | 334 | 349 | 683
  Unknown or Not Reported | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 8 | 21
  Asian | 172 | 173 | 345
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 5 | 8 | 13
  White | 173 | 172 | 345
  More than one race | 12 | 10 | 22
  Unknown or Not Reported | 18 | 28 | 46
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) or 2 (Ambulatory but unable to work). The number of participants with missing ECOG performance status is indicated for each treatment arm.
  Participants
    ECOG = 0 | 267 | 271 | 538
    ECOG = 1 | 127 | 126 | 253
    ECOG = 2 | 1 | 0 | 1
    Missing | 0 | 2 | 2
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in this study was stratified by geographic region of the enrolling site (Asia without Japan versus Japan and Western regions).
  Participants
    Asia without Japan | 121 | 123 | 244
    Japan and Western regions | 274 | 276 | 550

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from the date of the first documentation of disease progression, as determined by blinded independent central review (BICR) per RECIST 1.1 or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: Up to approximately 41 months
Population: The analysis population consisted of all randomized participants. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Months | 8.2 [6.3 to 8.3] | 8.1 [6.3 to 8.3]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Hazard Ratio (HR) = 0.834, 95% CI 2-sided [0.712 to 0.978] — Based on Cox model with Efron's method of tie handling with treatment as a covariate stratified by geographic region, MPVI or extrahepatic spread or both, AFP and ECOG PS

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization until death from any cause
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Months | 21.2 [19.0 to 23.6] | 19.0 [17.2 to 21.7]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Superiority; p = 0.0227, Log Rank; Onesided p-value based on logrank test stratified by geographic region, portal vein invasion/extrahepatic spread/both AFP status,ECOG status; Hazard Ratio (HR) = 0.840, 95% CI 2-sided [0.708 to 0.997] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 as assessed by BICR. RECIST 1.1 has been modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Percentage of Participants | 26.1 [21.8 to 30.7] | 17.5 [13.9 to 21.6]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Difference in percentage = 8.5, 95% CI 2-sided [2.8 to 14.2] — Based on Miettinen & Nurminen method stratified by geographic region, MPVI or extrahepatic spread or both, AFP and ECOG PS

4. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR was determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR, per RECIST 1.1 as assessed by BICR, until the first documented disease progression or death due to any cause, whichever occurred first. RECIST 1.1 has been modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 41 months
Population: The analysis population consisted of all randomized participants. Participants were analyzed based on the population of responders (participants that achieved complete or partial response).
Measure: Median (Full Range); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 103 | 70
Months | 4.1 [1.3 to 25.3] | 4.0 [0.3 to 18.6]

5. Secondary Outcome: Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DCR was defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD) per RECIST 1.1 as assessed by BICR. SD must be achieved at ≥6 weeks after randomization to be considered best overall response. RECIST 1.1 has been modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Percentage of Participants | 81.3 [77.1 to 85.0] | 78.4 [74.1 to 82.4]

6. Secondary Outcome: Time to Disease Progression (TTP) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by BICR. RECIST 1.1 was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ were followed.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Months | 8.3 [8.1 to 10.3] | 8.2 [7.0 to 8.4]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.93] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Progression-free Survival (PFS) Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: PFS was defined as the time from the first dose of study intervention to the first documented progressive disease (PD) per mRECIST by BICR or death due to any cause, whichever occurred first. mRECIST for HCC allowed evaluation of treatment effects that were not reflected in simple total size changes of lesions. Per mRECIST, PD was defined as an increase of at least 20% in the sum of diameters (SODs) of viable (enhancing) target lesions, taking as reference the smallest SODs of viable (enhancing) target lesions recorded since the treatment started.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Months | 8.4 [8.2 to 10.2] | 8.1 [6.5 to 8.3]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.68 to 0.94] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: ORR wass defined as the percentage of participants who have a confirmed complete response (CR: disappearance of any intratumoral arterial enhancement in all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of viable [enhancement in the arterial phase] target lesions, taking as reference the baseline sum of the diameters of target lesions) per mRECIST as assessed by BICR. mRECIST for hepatocellular carcinoma evaluates lesions within the liver parenchyma showing increased contrast enhancement in the arterial phase. A maximum of 10 target lesions and a maximum of 5 target lesions per organ were followed.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Percentage of Participants | 40.8 [35.9 to 45.8] | 34.1 [29.4 to 39.0]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Difference in percentage = 6.7, 95% CI 2-sided [0.0 to 13.4] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Duration of Response (DOR) Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: DOR was determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR, per mRECIST as assessed by BICR, until the first documented disease progression or death due to any cause, whichever occurs first. mRECIST for hepatocellular carcinoma evaluates lesions within the liver parenchyma showing increased contrast enhancement in the arterial phase. A maximum of 10 target lesions and a maximum of 5 target lesions per organ were followed.
Time Frame: Up to approximately 41 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment. Participants were analyzed based on the population of responders (participants that achieved complete or partial response).
Measure: Median (Full Range); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 151 | 136
Months | 2.1 [1.2 to 16.6] | 2.1 [0.2 to 14.5]

10. Secondary Outcome: Disease Control Rate (DCR) Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: DCR was defined as the percentage of participants who have a best overall response of CR, PR, or SD per mRECIST as assessed by BICR. mRECIST for hepatocellular carcinoma evaluates lesions within the liver parenchyma showing increased contrast enhancement in the arterial phase. SD must be achieved at ≥6 weeks after randomization to be considered best overall response. A maximum of 10 target lesions and a maximum of 5 target lesions per organ were followed.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Percentage of Participants | 84.3 [80.3 to 87.7] | 83.2 [79.2 to 86.7]

11. Secondary Outcome: Time to Disease Progression (TTP) Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: TTP was defined as the time from randomization to the first documented disease progression per mRECIST as assessed by BICR. mRECIST for hepatocellular carcinoma evaluates lesions within the liver parenchyma showing increased contrast enhancement in the arterial phase. A maximum of 10 target lesions and a maximum of 5 target lesions per organ were followed.
Time Frame: Up to approximately 41 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 399
Months | 10.4 [8.5 to 11.7] | 8.3 [8.1 to 8.9]
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs Lenvatinib + Placebo; Test type: Other — Descriptive assessment; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.61 to 0.88] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: Number of participants who experienced an AE defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study treatment
Time Frame: Up to approximately 68 months
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 395
Participants | 394 | 392

13. Secondary Outcome: Number of Participants Who Experienced an Serious Adverse Event (SAE)
Description: Number of participants who experienced a SAE defined as an AE that resulted in death, was life threatening, resulting in persistent or significant disability or incapacity, resulting in or prolonged a hospitalization, was a congenital anomaly or birth defect, was a cancer, was associated with an overdose, or was another important medical event
Time Frame: Up to approximately 68 months
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 395
Participants | 185 | 159

14. Secondary Outcome: Number of Participants Who Experienced an Immune-related Adverse Event (irAE) of Clinical Interest
Description: Number of participants who experienced an AE representing an immunologic etiology and considered to be causally related to drug exposure
Time Frame: Up to approximately 41 months
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 395
Participants | 210 | 184

15. Secondary Outcome: Number of Participants Who Experienced an Hepatic Event of Clinical Interest (HECI)
Description: Number of participants who experienced a hepatic ECI not due to disease progression as judged by the investigator.
Time Frame: Up to approximately 68 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 395
Participants | 71 | 77

16. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: Number of participants who discontinued study treatment due to an AE
Time Frame: Up to approximately 68 months
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
Number analyzed (Participants) | 395 | 395
Participants | 51 | 41

ADVERSE EVENTS:
Time Frame: Up to ~ 68 months
Description: All-cause mortality includes all randomized participants. Safety includes participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Lenvatinib + Pembrolizumab | Lenvatinib + Placebo
All-Cause Mortality (participants affected / at risk) | 314/395 | 352/399
Serious Adverse Events (participants affected / at risk) | 185/395 | 159/395
Other Adverse Events (participants affected / at risk) | 390/395 | 388/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=395) | Lenvatinib + Placebo (N=395)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (5) | 10 (10)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation, obstructive (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (5)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (5)
Varices oesophageal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 5 (5) | 3 (3)
Drowning (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 7 (8) | 0 (0)
Hyperthermia malignant (General disorders) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 4 (5)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (6)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 4 (5) | 8 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 3 (3)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 2 (3) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Biliary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (2) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pleurisy bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 7 (7)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (5) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1)
False positive investigation result (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 21 (27) | 11 (12)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Scrotal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive emergency (Vascular disorders) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=395) | Lenvatinib + Placebo (N=395)
Anaemia (Blood and lymphatic system disorders) | 51 (61) | 64 (88)
Neutropenia (Blood and lymphatic system disorders) | 19 (54) | 22 (38)
Hyperthyroidism (Endocrine disorders) | 31 (32) | 15 (16)
Hypothyroidism (Endocrine disorders) | 167 (207) | 159 (202)
Abdominal distension (Gastrointestinal disorders) | 27 (33) | 18 (20)
Abdominal pain (Gastrointestinal disorders) | 74 (88) | 74 (91)
Abdominal pain upper (Gastrointestinal disorders) | 46 (52) | 40 (53)
Ascites (Gastrointestinal disorders) | 28 (35) | 29 (34)
Constipation (Gastrointestinal disorders) | 67 (81) | 73 (81)
Diarrhoea (Gastrointestinal disorders) | 187 (359) | 167 (352)
Dry mouth (Gastrointestinal disorders) | 20 (20) | 14 (14)
Dyspepsia (Gastrointestinal disorders) | 33 (41) | 14 (18)
Nausea (Gastrointestinal disorders) | 89 (123) | 82 (120)
Stomatitis (Gastrointestinal disorders) | 41 (55) | 35 (47)
Toothache (Gastrointestinal disorders) | 24 (28) | 18 (23)
Vomiting (Gastrointestinal disorders) | 54 (93) | 61 (93)
Asthenia (General disorders) | 73 (90) | 61 (85)
Fatigue (General disorders) | 126 (148) | 98 (124)
Malaise (General disorders) | 20 (24) | 30 (35)
Mucosal inflammation (General disorders) | 25 (30) | 19 (25)
Oedema peripheral (General disorders) | 63 (86) | 54 (68)
Pyrexia (General disorders) | 48 (60) | 45 (66)
Upper respiratory tract infection (Infections and infestations) | 20 (27) | 14 (16)
Urinary tract infection (Infections and infestations) | 35 (48) | 42 (65)
Alanine aminotransferase increased (Investigations) | 93 (162) | 89 (155)
Amylase increased (Investigations) | 40 (64) | 18 (30)
Aspartate aminotransferase increased (Investigations) | 117 (195) | 105 (179)
Blood alkaline phosphatase increased (Investigations) | 50 (64) | 35 (54)
Blood bilirubin increased (Investigations) | 101 (222) | 108 (216)
Blood creatinine increased (Investigations) | 39 (60) | 25 (41)
Gamma-glutamyltransferase increased (Investigations) | 65 (78) | 56 (72)
Lipase increased (Investigations) | 57 (79) | 37 (59)
Neutrophil count decreased (Investigations) | 34 (73) | 39 (85)
Platelet count decreased (Investigations) | 101 (170) | 110 (198)
Weight decreased (Investigations) | 121 (139) | 90 (105)
White blood cell count decreased (Investigations) | 29 (75) | 45 (105)
Decreased appetite (Metabolism and nutrition disorders) | 146 (183) | 120 (167)
Hyperglycaemia (Metabolism and nutrition disorders) | 24 (33) | 25 (46)
Hyperkalaemia (Metabolism and nutrition disorders) | 14 (22) | 20 (26)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 24 (51) | 31 (64)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 62 (85) | 61 (99)
Hypokalaemia (Metabolism and nutrition disorders) | 39 (75) | 36 (60)
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 (46) | 28 (56)
Hyponatraemia (Metabolism and nutrition disorders) | 43 (69) | 39 (64)
Hypophosphataemia (Metabolism and nutrition disorders) | 19 (24) | 23 (43)
Arthralgia (Musculoskeletal and connective tissue disorders) | 89 (114) | 77 (93)
Back pain (Musculoskeletal and connective tissue disorders) | 60 (72) | 43 (49)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (27) | 14 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (22) | 23 (27)
Dizziness (Nervous system disorders) | 26 (30) | 28 (30)
Dysgeusia (Nervous system disorders) | 22 (26) | 19 (21)
Headache (Nervous system disorders) | 51 (67) | 43 (58)
Insomnia (Psychiatric disorders) | 35 (40) | 43 (49)
Haematuria (Renal and urinary disorders) | 27 (43) | 24 (55)
Proteinuria (Renal and urinary disorders) | 136 (280) | 153 (268)
Cough (Respiratory, thoracic and mediastinal disorders) | 55 (66) | 43 (49)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 83 (94) | 79 (92)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (47) | 24 (32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 29 (42)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 15 (17)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 133 (155) | 125 (141)
Pruritus (Skin and subcutaneous tissue disorders) | 67 (79) | 44 (57)
Rash (Skin and subcutaneous tissue disorders) | 63 (79) | 35 (46)
Hypertension (Vascular disorders) | 180 (248) | 200 (258)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT03713593/Prot_SAP_001.pdf